CLINICAL TRIAL: NCT02542319
Title: The Effect of Oral Magnesium Supplementation on Vascular Calcification in Chronic Kidney Disease - A Randomized Clinical Trial
Brief Title: Effect of Oral Magnesium on Vascular Calcification in Chronic Kidney Disease
Acronym: MagiCal-CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MagiCal-CKD
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2018-06

CONDITIONS: Chronic Kidney Disease; Vascular Calcification; Uremic Osteodystrophy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vascular Calcification

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium (Experimental): Oral Magnesium Hydroxide (Mablet 360 mg) twice daily for 12 months.
  Interventions: Dietary Supplement: Mablet 360 mg
- Placebo (Placebo Comparator): Matching placebo tablets twice daily for 12 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mablet 360 mg
  Arms: Magnesium
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Randomized placebo-controlled double-blinded interventional trial to investigate the effect of oral magnesium supplementation on vascular calcification in subjects with chronic kidney disease. We hypothesize that oral magnesium supplementation will reduce vascular calcification in subjects with chronic kidney disease while not decreasing bone mineral density.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is associated with increase cardiovascular morbidity and mortality independent of traditional cardiovascular risk factors due to increased vascular calcification. Epidemiological and experimental data suggest that hypermagnesemia and magnesium supplementation reduce vascular calcification in CKD by increasing calcium/phosphate solubility in serum, by inhibiting calcium influx into vascular smooth muscle cells (VSMC), by inhibiting intracellular pro-calcification enzymes in VSMC and by increasing activity of intracellular anti-calcification enzymes in VSMC. However, there have been concerns that any anti-calcification effect of magnesium might also reduce bone mineral density, in which case there might be an increased risk of bone fractures associated with magnesium supplementation in CKD. We wish to conduct a randomized placebo-controlled double-blinded interventional trial to examine whether oral magnesium supplementation will reduce vascular calcification in subjects with CKD while not decreasing bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate between 45 and 15 mL/min for > 3 months (i.e. CKD stage 3b-4).
* Serum total magnesium < 0,82 mmol/L and serum phosphate > 1,15 mmol/L on average of previous measurements.

or Serum total magnesium < 0,92 mmol/L and serum phosphate > 1,30 mmol/L on average of previous measurements.

* Life expectancy > 1 year.
* Expected time until initiation of dialysis or transplantation > 1 year.
* Women of childbearing age must be actively using contraceptive therapy (p-pills, estrogen depots or intrauterine device) as well as have a negative pregnancy test.
* Written informed consent.

Exclusion Criteria:

* Current hemodialysis or peritoneal dialysis treatment.
* Kidney donor recipient.
* Previous coronary artery bypass graft (CABG).
* Parathyroid hormone > 600 ρmol/L.
* Previous parathyroidectomy.
* Current treatment with magnesium containing medication or supplements.
* Any condition impairing magnesium absorption from the gastrointestinal tract (e.g. short bowel syndrome, chronic pancreatitis).
* Active malignancy (basal or squamous cell skin carcinoma, localized prostate cancer and cancer with no signs of reoccurrence after 5 years are exempt from this).
* Other diseases or conditions, which, in the opinion of the site investigator, would prevent participation in or completion of trial.
* Pregnancy or breastfeeding.
* Allergy towards contents of interventional medication.
* Participation in other interventional trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-11; Primary Completion 2020-11 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Calcification (CAC) score | 12 months
  Agatston score assessed by CT scan.

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) | 12 months
  BMD assessed by quantitative CT.
Pulse Wave Velocity | 12 months.
Serum Calcification Propensity | 12 months.
  Serum calcification propensity assessed by T50 analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Iain O Bressendorff, MD, PhD, Principal Investigator — Nordsjaellands Hospital
Locations (3):
- Denmark (2):
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
- Akershus Universitetssykehus, Lørenskog, Norway

REFERENCES:
- [Derived] Bressendorff I, Hansen D, Schou M, Kragelund C, Svensson M, Hashemi B, Kristensen T, Vrist MH, Borg R, Tougaard B, Borg K, Hjortkjaer HO, Kristiansen CH, Carlson N, Nasiri M, Ashraf H, Pasch A, Brandi L. The Effect of Magnesium Supplementation on Vascular Calcification in CKD: A Randomized Clinical Trial (MAGiCAL-CKD). J Am Soc Nephrol. 2023 May 1;34(5):886-894. doi: 10.1681/ASN.0000000000000092. Epub 2023 Feb 2. PMID 36749131
- [Derived] Bressendorff I, Hansen D, Schou M, Kragelund C, Brandi L. The effect of magnesium supplementation on vascular calcification in chronic kidney disease-a randomised clinical trial (MAGiCAL-CKD): essential study design and rationale. BMJ Open. 2017 Jun 23;7(6):e016795. doi: 10.1136/bmjopen-2017-016795. PMID 28645983